CLINICAL TRIAL: NCT06873113
Title: Blood Flow Restriction Training for Subacromial Pain: A Pilot Randomized Controlled Trial
Brief Title: BFRT for Subacromial Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB202302184; R21AR082588-01A1 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Pain
Keywords: blood flow restriction training; BFRT; BFR; exercise; subacromial pain; rotator cuff tendinopathy; subacromial impingement; rotator cuff related shoulder pain
MeSH Terms: conditions — Shoulder Pain; Motor Activity; Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active BFRT (Experimental)
  Interventions: Device: Active BFRT; Behavioral: Strengthening Exercises with BFRT; Behavioral: Skilled Physical Therapy Care
- Sham BFRT (Sham Comparator)
  Interventions: Device: Sham BFRT; Behavioral: Strengthening Exercises with BFRT; Behavioral: Skilled Physical Therapy Care

INTERVENTIONS:
Device: Active BFRT — The BFR device is applied unilaterally on participants involved upper extremity. The BFR device maintains 50% of participants limb occlusion pressure for the duration of each strengthening exercise.
  Arms: Active BFRT
Device: Sham BFRT — The BFR device is applied unilaterally on participants involved upper extremity. The BFR device maintains a pressure of 20mmHg for the duration of each strengthening exercise.
  Arms: Sham BFRT
Behavioral: Strengthening Exercises with BFRT — Participants perform 4 strengthening exercises while using the BFR device: seated scapular plane elevation, prone horizontal abduction, side-lying external rotation, and prone scapular plane elevation. Each exercise is performed unilaterally. Participants perform 1 set of 30 repetitions followed by 3 sets of 15 repetitions (4 total sets, 75 total repetitions). Participants are given 30 seconds rest between sets and 2 minutes of rest between strengthening exercises. Selected resistance for each strengthening exercise is equal to 20% of the participant's maximal force production as measured by handheld dynamometry. Resistance is adjusted weekly.
Behavioral: Skilled Physical Therapy Care — Participants perform non-strengthening interventions as part of skilled physical therapy care. Non-strengthening interventions include an upper arm ergometer for warm-up, active assisted range of motion of the shoulder, shoulder stretching, shoulder joint mobilizations, and cryotherapy. Non-strengthening interventions are prescribed at the discretion of the treating physical therapist. Participants are enrolled in physical therapy for a minimum of 4 weeks. After 4 weeks, the treating physical therapist can discharge a participant based on their progress in meeting their rehabilitation goals. Participants discharged from skilled physical therapy care will continue to complete strengthening exercises with BFRT until the end of the trial period (8 weeks).

SUMMARY:
The goal of this pilot clinical trial is to learn if blood flow restriction training is safe and feasible in patients with subacromial pain. The main questions the investigators aim to answer are:

* What problems do participants with shoulder pain encounter when training with blood flow restriction?
* Is it feasible to apply blood flow restriction training as part of a physical therapy intervention?
* What are some preliminary effects of blood flow restriction training on the recovery of shoulder function and strength?

The investigators will compare active blood flow restriction training to sham (an inactive procedure designed to mimic the active training as closely as possible).

Participants will:

* Visit the clinic for physical therapy visits and exercise with blood flow restriction training for up to 8 weeks
* Visit the clinic for tests before starting the treatment, during the treatment (4 weeks), and after the end of the treatment (8 and 26 weeks).

ELIGIBILITY:
Inclusion criteria

* Between 18 and 50 years of age
* Unilateral pain in the anterolateral shoulder
* Self-reported shoulder function of ≤7 (10, full function)
* At least 90° of active shoulder elevation
* 3 out of 5 positive tests to define subacromial pain.

Exclusion Criteria (general):

* history of shoulder fracture, frozen shoulder, or shoulder surgery
* primary complaint of shoulder instability/dislocation
* history of cardiovascular, neurologic, and pulmonary conditions that would impair the subject's ability to participate in physical therapy
* active treatment for cancer
* uncontrolled diabetes
* uncontrolled high blood pressure
* corticosteroid injection at the shoulder within 6 weeks
* imaging evidence of rotator cuff tears
* pregnancy

Exclusion criteria (Blood flow restriction training specific)

* contraindications to BFRT (sickle cell anemia, deep vein thrombosis, peripheral circulatory diseases)
* taking anticoagulant or antiplatelet drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Monthly report from beginning to completion of recruitment (anticipated 2 years)
  Record the number of individuals a) approached, b) screened, c) qualified, and d) willing to participate. The reasons for participants who do not qualify or refuse to participate will be recorded.
Intervention feasibility | Weekly record from enrollment to the end of treatment at 8 weeks.
  The interventionist team will complete standardized notes of the intervention, which will be reviewed weekly to document adherence and protocol fidelity and for early identification of intervention deviations. Outcomes include the number of patients a) completing at least 80% of the assigned BFRT visits, b) requesting to stop BFRT within a session, c) requesting to withdraw from the intervention, and d) requesting to switch intervention arms. The last number is a proxy for patients who do not accept randomization results.

SECONDARY OUTCOMES:
Retention | Weekly record from enrollment to 26 weeks (end of the trial).
  Identify the number of dropouts and reasons impacting participation in follow-up visits.
Intervention safety | Weekly record from enrollment to 26 weeks (end of the trial).
  Monitor the occurrance of severe adverse events and exercise-related adverse events.
Participants masking feasibility | At 8 weeks
  At the primary endpoint, participants will be asked to guess the treatment allocation to evaluate participant masking feasibility.
Patient acceptability | At 8 weeks
  A guided interview using Likert scale-type and open-ended questions will be conducted to gather participant feedback on trial and intervention procedures. An electronic copy of this questionnaire will be sent to patients who withdraw/stop showing up to understand whether trial or intervention procedures impact patient retention.
Range of motion | From enrollment to 4 weeks, 8 weeks and 6 months
  The investigators will measure range of motion using an inclinometer or goniometer. The investigators will measure shoulder elevation in the scapular plane, external rotation, and internal rotation. The investigators will also measure coronal, axial, and sagittal rotation of the scapula during shoulder elevation in the scapular plane.
Strength | From enrollment to 4 weeks, 8 weeks and 6 months
  The investigators will measure shoulder elevation in the scapular plane and external rotation strength using a handheld dynamometer.
Timed Functional Arm and Shoulder Test (TFAST) | From enrollment to 4 weeks, 8 weeks and 6 months
  It includes three tasks: an internal/external rotation task (duration 30s), an outward circular motion task (duration 30s), and a gallon-lift task at the height of a standard counter (duration 30s). In each task, participants repeat movements as fast as possible.
Supraspinatus and infraspinatus muscle cross-sectional area | From enrollment to 4 weeks, 8 weeks and 6 months
  The investigators will use ultrasound to take pictures of the supraspinatus and infraspinatus muscles. This outcome represents a marker of hypertrophy, a potential mechanism of strengthening.
Supraspinatus tendon morphology | From enrollment to 4 weeks, 8 weeks and 6 months
  The investigators will use ultrasound to take pictures of the supraspinatus tendons. Established ultrasound procedures will be used to measure supraspinatus tendon thickness.
Supraspinatus tendon elastography | From enrollment to 4 weeks, 8 weeks and 6 months
  Ultrasound will be used to take pictures of the supraspinatus tendons. The investigators will set the ultrasound parameters to elastography, allowing non-invasive measurement of tendon stiffness and elasticity.
Pennsylvania Shoulder Score (PENN) | From enrollment to 4 weeks, 8 weeks and 6 months
  The PENN is a valid and reliable self-reported questionnaire for patients with shoulder pain.
Global rating of change (GROC) | At 4 weeks, 8 weeks and 6 months
  The GROC is a rating scale that quantifies participants' improvement or deterioration of symptoms over time. Changes will be measured using a 15-points Likert scale (-7, a very great deal worse to 7, a very great deal better, with 0 indicating no changes).
Patient specific functional scale (PSFS) | From enrollment to 4 weeks, 8 weeks and 6 months
  The PSFS asks patients to rate their difficulty performing three activities of their choice. It is advantageous because it asks patients to select the activities rather than providing pre-selected options.

OTHER OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | From enrollment to 4 weeks, 8 weeks and 6 months
  The WORC is a valid and reliable tool to assess quality of life in patients with shoulder pain. The tool contains a total of 21 Likert-type questions in five different domains (Physical symptoms, Sports/Recreation/Work/Lifestyle/Emotions)
Brief Pain Inventory (BPI) | From enrollment to 4 weeks, 8 weeks and 6 months
  The BPI is a reliable, primary pain recovery measure used in clinical trials of patients with shoulder pain. It measures pain across three domains (average, best, and worst).
Patient Acceptable Symptoms State (PASS) | At 8 weeks and 6 months
  The PASS is a rating scale that quantifies participants' satisfaction with their current level of function in the context of clinical care.
Pressure pain sensitivity | From enrollment to 4 weeks, 8 weeks and 6 months
  The investigators will apply pressure at a constant rate using a computerized pressure algometer with a 1 cm diameter rubber tip at the shoulder and the lower limb.
Quick Disability of the Arm and Shoulder (Q-DASH) | From enrollment to 4 weeks, 8 weeks and 6 months
  The Q-DASH evaluates upper extremity disability while monitoring change or function over time. This assessment consists of 11 questions (3 items related to symptoms and 8 items related to functional tasks). Reliability and validity have been established for this scale.
Infraspinatus tendon morphology | From enrollment to 4 weeks, 8 weeks and 6 months
  The investigators will use ultrasound to take pictures of the infraspinatus tendons. Established ultrasound procedures will be used to measure infraspinatus tendon thickness.
Infraspinatus tendon elastography | From enrollment to 4 weeks, 8 weeks and 6 months
  Ultrasound will be used to take pictures of the infraspinatus tendons. The investigators will set the ultrasound parameters to elastography, allowing non-invasive measurement of tendon stiffness and elasticity.
Optimal Screening for Prediction of Referral and Outcome (OSPRO) | From enrollment to 4 weeks, 8 weeks and 6 months
  The OSPRO is a concise, multidimensional 10-item yellow flag assessment tool that estimates 11 total questionnaire scores indicating elevated vulnerability and decreased resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Study protocol & statistical analysis plan: A manuscript describing the study protocol and statistical analysis plan will be submitted for publication within the first year of starting the clinical trial.
  Clinical study report and analytic code: Individual data and analytic code will be made available after the publication of the primary results of this trial.
Access Criteria: Study protocol and statistical analysis plan: The manuscript will be published as open access.
  Clinical study report and analytic code: Data will be shared on NIH/NIAMS approvved data repository (i.e., Dataverse). Access will follow repository guidelines.